CLINICAL TRIAL: NCT06627647
Title: A Phase III, Randomized, Double-blind, Multicenter, Global Study of Rilvegostomig or Pembrolizumab in Combination With Platinum-based Chemotherapy for the First-line Treatment of Patients With Metastatic Non-squamous Non-small Cell Lung Cancer Whose Tumors Express PD-L1 (ARTEMIDE-Lung03)
Brief Title: A Global Phase III Study of Rilvegostomig or Pembrolizumab Plus Chemotherapy for First-Line Treatment of Metastatic Non-squamous NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D702FC00001; 2024-515008-38-00 (Other: CTIS ID)
Record Dates: First submitted 2024-10-03; First posted 2024-10-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
Keywords: ARTEMIDE-Lung03; Rilvegostomig (AZD2936); Non-squamous non-small cell lung cancer (NSCLC); Bi-specific antibody; T-cell immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domain (TIGIT); EGFR, ALK and ROS1 testing; Programmed cell death protein (PD-L1); Pembrolizumab; Carboplatin; Cisplatin; Pemetrexed
MeSH Terms: interventions — pembrolizumab; Carboplatin; Cisplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Arm A: Rilvegostomig in combination with platinum-based doublet chemotherapy followed by rilvegostomig monotherapy plus pemetrexed in maintenance.
  Arm B: Pembrolizumab in combination with platinum-based doublet chemotherapy followed by pembrolizumab monotherapy plus pemetrexed in maintenance.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Rilvegostomig in combination with platinum-based doublet chemotherapy followed by rilvegostomig monotherapy plus pemetrexed in maintenance.
  Interventions: Drug: Rilvegostomig; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed
- Arm B (Active Comparator): Pembrolizumab in combination with platinum-based doublet chemotherapy followed by pembrolizumab monotherapy plus pemetrexed in maintenance.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Rilvegostomig — Administered as one intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: AZD2936
  Arms: Arm A
Drug: Pembrolizumab — Administered as one intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: Keytruda
  Arms: Arm B
Drug: Carboplatin — Administered as one intravenously (IV) on Day 1 of each 21-day cycle up to 4 cycles
Drug: Cisplatin — Administered as one intravenously (IV) on Day 1 of each 21-day cycle up to 4 cycles
Drug: Pemetrexed — Administered as one intravenously (IV) on Day 1 of each 21-day cycle

SUMMARY:
The purpose of ARTEMIDE-Lung03 is to evaluate the efficacy and safety of rilvegostomig compared to pembrolizumab, both in combination with platinum-based doublet chemotherapy, as a first-line treatment of patients with non-squamous mNSCLC whose tumors express PD-L1.

DETAILED DESCRIPTION:
This is a Phase III, two-arm, randomized, double-blind, global, multicenter study assessing the efficacy and safety of rilvegostomig compared to pembrolizumab, both in combination with platinum-based doublet chemotherapy, as a 1L treatment for patients with non-squamous mNSCLC whose tumors express PD-L1 (TC ≥ 1%).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented non-squamous NSCLC.
* Stage IV mNSCLC (based on the American Joint Committee on Cancer Edition 8) not amenable to curative treatment.
* Absence of sensitizing EGFR mutations (including, but not limited to, exon 19 deletion and exon 21 L858R, exon 21 L861Q, exon 18 G719X, and exon 20 S768I mutations) and ALK and ROS1 rearrangements.
* Absence of documented tumor genomic mutation results from tests conducted as part of standard local practice in any other actionable driver oncogenes for which there are locally approved targeted 1L therapies.
* Provision of acceptable tumor sample, to confirm tumor PD-L1 expression TC ≥ 1%.
* At least one lesion not previously irradiated that qualifies as a RECIST 1.1 TL at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with CT or MRI and is suitable for accurate repeated measurements.
* Adequate organ and bone marrow function

Exclusion Criteria:

* Presence of small cell and neuroendocrine histology components.
* Brain metastases unless asymptomatic, stable, and not requiring steroids or anticonvulsants for at least 7 days prior to randomization. A minimum of 2 weeks must have elapsed between the end of local therapy (brain radiotherapy or surgery) and randomization. Participants must have recovered from the acute toxic effect of radiotherapy (eg, dizziness and signs of increased intracranial pressure) or surgery prior to randomization.
* Any prior systemic therapy received for advanced or mNSCLC. Prior systemic therapy in the neoadjuvant or adjuvant setting and/or definitive radio- or chemoradiotherapy for early-stage disease are allowed, provided that recurrence or progression has occurred > 12 months after the end of treatment.
* Any prior exposure to an anti-TIGIT therapy or any other anticancer therapy targeting immune-regulatory receptors or mechanisms.
* Any prior treatment with an anti-PD-1 or anti-PD-L1 agent.
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence.
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment.
* Active primary immunodeficiency/active infectious disease(s).
* Active tuberculosis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2029-05-10 (Estimated); Study Completion 2030-03-25 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Progression-free survival (PFS) | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1, or death due to any cause (in the absence of progression).

SECONDARY OUTCOMES:
Landmark overall survival (OS) rates | Up to approximately 5 years
  OS is defined as the time from randomization until the date of death due to any cause.
Landmark progression-free survival (PFS) rates | Up to approximately 5 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1, or death due to any cause (in the absence of progression).
Time to second progression or death (PFS2) | Up to approximately 5 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial progression event), after the start of the first subsequent therapy, or death from any cause, whichever occurs first. The date of the second progression will be recorded by the investigator in the eCRF and defined according to local standard clinical practice.
Overall response rate (ORR) | Up to approximately 5 years
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, using RECIST 1.1.
Duration of response (DoR) | Up to approximately 5 years
  DoR is defined as the time from the date of first documented response until the date of documented progression using RECIST 1.1 or death due to any cause (in the absence of progression).
Pharmacokinetic (PK) of rilvegostomig | Up to approximately 5 years
  Concentration of rilvegostomig in serum
Immunogenicity of rilvegostomig | Up to approximately 5 years
  Presence of antidrug antibodies (ADAs), titer, and neutralizing antibodies for rilvegostomig
Patient-reported physical functioning | Up to approximately 5 years
  Proportion of participants with maintained or improved physical functioning as measured by PROMIS PF-SF 8c - 7 day at each time point.
Patient-reported global health status (GHS)/quality of life (QoL) | Up to approximately 5 years
  TTD of GHS/QoL as measured by the EORTC IL172. TTD is defined as time from randomization to the date of first deterioration. Deterioration is defined as a worsening change from baseline that reaches a clinically meaningful change threshold.
Patient-reported lung cancer symptoms of non-small cell lung cancer (NSCLC) | Up to approximately 5 years
  TTD in pulmonary symptoms as measured by the NSCLC-SAQ. TTD is defined as time from randomization to the date of first deterioration.

CONTACTS AND LOCATIONS:
Locations (249):
- United States (74):
  - Research Site, Mobile, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Loma Linda, California
  - Research Site, Redlands, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Rosa, California
  - Research Site, Walnut Creek, California
  - Research Site, Lone Tree, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, West Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Bay Pines, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Decatur, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Quincy, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Waterloo, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, South Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Camden, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Westbury, New York
  - Research Site, Canton, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Pierre, South Dakota
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Kingwood, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Palestine, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Silverdale, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, La Crosse, Wisconsin
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Plata
  - Research Site, Pilar
  - Research Site, Rosario
- Australia (4):
  - Research Site, Darlinghurst
  - Research Site, Hyde Park
  - Research Site, Southport
  - Research Site, Wollongong
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Kortrijk
  - Research Site, Ottignies
  - Research Site, Sint-Niklaas
- Brazil (8):
  - Research Site, Ijuí
  - Research Site, Londrina
  - Research Site, Passo Fundo
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Vitória
- Canada (7):
  - Research Site, Saint John, New Brunswick
  - Research Site, Sydney, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
- China (22):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Jingzhou
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiangyang
  - Research Site, Zhengzhou
- France (8):
  - Research Site, Avignon
  - Research Site, La Rochelle
  - Research Site, Lyon
  - Research Site, Nîmes
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Toulon
- Germany (20):
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt
  - Research Site, Gauting
  - Research Site, Giessen
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Hemer
  - Research Site, Homburg
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Krefeld
  - Research Site, Minden
  - Research Site, Moers
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Würzburg
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- India (8):
  - Research Site, Calicut
  - Research Site, Delhi
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Varanasi
- Italy (4):
  - Research Site, Florence
  - Research Site, Monza
  - Research Site, Peschiera del Garda
  - Research Site, Rome
- Japan (22):
  - Research Site, Amagasaki-shi
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Kawagoe-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsusaka-shi
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Saitama-shi
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Takaoka-shi
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Petaling Jaya
- Netherlands (5):
  - Research Site, Alkmaar
  - Research Site, Ede
  - Research Site, Groningen
  - Research Site, Leidschendam
  - Research Site, Veldhoven
- Research Site, Lima, Peru
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Biała Podlaska
  - Research Site, Bydgoszcz
  - Research Site, Bystra
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- South Korea (3):
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
  - Research Site, Songpa-gu
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Castellon
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Nakhon Ratchasima
  - Research Site, Songkhla
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Edirne
  - Research Site, Izmir
  - Research Site, Seyhan
- United Kingdom (9):
  - Research Site, Aberdeen
  - Research Site, Cambridge
  - Research Site, Edinburgh
  - Research Site, Exeter
  - Research Site, Greater London
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Torquay
- Vietnam (4):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/